CLINICAL TRIAL: NCT00644748
Title: An Open, Multicenter Study on the Efficacy, Safety and Tolerability of Gabapentin, Titrated for Reaching an Effect for the Treatment of the Painful Diabetic Neuropathy
Brief Title: A Study on the Efficacy and Safety of Gabapentin in the Treatment of Patients With Painful Diabetic Neuropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A9451004
Record Dates: First submitted 2008-03-25; First posted 2008-03-27 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2008-10

CONDITIONS: Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gabapentin group (Experimental)
  Interventions: Drug: gabapentin

INTERVENTIONS:
Drug: gabapentin — Gabapentin oral capsules:
  Week 0: Day 1: 300 mg; Day 2: 600 mg (2 doses of 300 mg); Day 3: 900 mg (3 doses of 300 mg), maintained until the end of the week; After this point, the total daily dose was divided in 3 equal doses. Week 1: Day 1: 1200 mg; Day 2 to 7: 1800 mg Week 2: Day 1: 2100 mg; Day 2 to 7: 2400 mg Week 3: Day 1: 2700 mg; Day 2 to 7: 3600 mg Weeks 4 to 11: 3600 mg

SUMMARY:
The purpose of this study was to evaluate the efficacy, safety, and tolerability of gabapentin for the treatment of patients with painful diabetic neuropathy. The quality of life of all treated patients was also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable Diabetes Mellitus 1 or 2
* Clinical diagnosis of distal symmetric polyneuropathy with a minimum duration of 8 weeks
* No clinically significant motor deficits
* Pain described according to at least one of the following clinical manifestations: burning, cramps or twinges, thermal or mechanical alodinea

Exclusion Criteria:

* Treatment with any medication that may interfere with the assessment of gabapentin during the study or within 7 days of the adminstration of gabapentin
* Specific systemic diseases or other medical conditions that would interfere with the assessment of gabapentin therapeutic response or safety

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2003-05; Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline Mean Pain Score | Endpoint

SECONDARY OUTCOMES:
Change from baseline Mean Pain Score | Weekly
Proportion of responding patients | Endpoint
Change from baseline Mean Pain Interference with Sleep Score | Weekly and Endpoint
Change from baseline in the 5 sub-scores of the McGill Reduced Pain Questionnaire: the sensory score, the affective score, the total score for pain descriptors, a visual analogue scale, and a scale of Present Pain Intensity | Endpoint
Global Change Impression from the Patient's Point of View | Endpoint
Change from baseline in quality of life | Endpoint
Global Change Impression from the Physician's Point of View | Endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- Brazil (8):
  - Pfizer Investigational Site, Fortaleza, Ceará
  - Pfizer Investigational Site, Taguatinga, Federal District
  - Pfizer Investigational Site, Belo Horizonte, Minas Gerais
  - Pfizer Investigational Site, Curitiba, Paraná
  - Pfizer Investigational Site, Recife, Pernambuco
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São Paulo, São Paulo
- Pfizer Investigational Site

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9451004&StudyName=A%20study%20on%20the%20efficacy%20and%20safety%20of%20gabapentin%20in%20the%20treatment%20of%20patients%20with%20painful%20diabetic%20neuropathy